CLINICAL TRIAL: NCT01169896
Title: Impact of Ventricular Pacing in Unselected ICD/CRT-D Patients
Acronym: FIRST
Status: Completed | Type: Observational
Sponsor: LivaNova (Industry)
Responsible Party: Sponsor
Other Study IDs: RTGX01
Record Dates: First submitted 2010-07-22; First posted 2010-07-26 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Ventricular Tachycardia; Ventricular Fibrillation
Keywords: Impact of ventricular pacing on the incidence of VT/VF episodes for each models
MeSH Terms: conditions — Tachycardia, Ventricular; Ventricular Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Observational study is evaluating Ventricular Tachycardia (VT)/Ventricular Fibrillation (VF) thérapies as a function of ventricular pacing

DETAILED DESCRIPTION:
This protocol consists in a non-interventional multi-centre, prospective study. The observational study will also answer the question of the impact of ventricular pacing on the outcome of patients implanted with ICD & CRT-D devices and how the ICD & CRT-D devices are used in clinical practice through two years follow-up.

ELIGIBILITY:
Main inclusion Criteria:

•Patient implanted (primo implantation or replacement) with an ICD (OVATIO VR 6250, DR 6550, CRT 6750 models, or any similar or higher range device, that includes specific diagnostic and therapeutic functionalities, mandatory to make homogeneous the collection of data)

Main exclusion Criteria:

* Presence of a contra-indication to the ICD therapy.
* Life expectancy less than 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: unselected ICD/CRT-D implanted patients
Sampling Method: Probability Sample
Enrollment: 616 (Actual)
Dates: Start 2007-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
VT/VF episodes according to ventricular pacing (> and <50%) | 2 years
  Device-based data

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Piot, MD, Principal Investigator — CCN St Denis
Locations (1):
- CCN, Saint-Denis, France